CLINICAL TRIAL: NCT05650658
Title: Cardiac Resynchronization Therapy Using His/Left Bundle Branch Pacing vs Biventricular Pacing With a Left Ventricular Epicardial Lead in Patients With Heart Failure (HF) With Left Ventricular Ejection Fraction (LVEF)≤50% and With Either a Wide QRS Complex (>130 ms) or With/Anticipated >40% Pacing Randomized Clinical Trial
Brief Title: Left vs Left Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Utah (Other); Virginia Commonwealth University (Other); Cleveland Clinic Florida (Other); East Carolina University (Other)
Responsible Party: Principal Investigator, Mihail Gabriel Chelu, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PLACER 2021C3- 24160
Record Dates: First submitted 2022-11-24; First posted 2022-12-14 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction; AV Block; LBBB; RBBB; Intraventricular Conduction Delay; Pacing-Induced Cardiomyopathy
MeSH Terms: conditions — Heart Failure; Atrioventricular Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- His/Left Bundle Branch Pacing (His/LBBP) (Active Comparator): Patients with LVEF≤35% at entry will receive a His/LBB defibrillator which includes implantation of three leads, an endocardial right atrial lead, an endocardial right ventricular ICD lead, and an endocardial His-bundle or left bundle branch pacing lead directly pacing the intrinsic conduction system.
  Patients with LVEF 36-50% at entry will receive His/LBB pacemaker which includes implantation of two leads, an endocardial right atrial lead, and an endocardial His-bundle or left bundle branch pacing lead directly pacing the intrinsic conduction system.
  Interventions: Device: His/LBBP
- Biventricular Pacing (BiVP) (Active Comparator): Patients with LVEF≤35% at entry will receive a BiV defibrillator which includes implantation of three leads, an endocardial right atrial lead, an endocardial right ventricular ICD lead, and and an epicardial left ventricular lead implanted in a branch of the coronary sinus.
  Patients with LVEF 36-50% at entry will receive BiV pacemaker which includes implantation of three leads, an endocardial right atrial lead, an endocardial right ventricular pacing lead, and and an epicardial left ventricular lead implanted in a branch of the coronary sinus.
  Interventions: Device: BiVP

INTERVENTIONS:
Device: His/LBBP — Pacing at the level His-Bundle or left bundle branch is used to correct the underlying conduction abnormality, resulting in a faster and more homogeneous activation of the heart pacing directly via the intrinsic conduction system of the heart accompanied by a right atrial endocardial lead and a right ventricular defibrillator endocardial lead for LVEF≤35% and by a right atrial endocardial lead for LVEF 36-50%.
  Arms: His/Left Bundle Branch Pacing (His/LBBP)
Device: BiVP — Biventricular pacing has been shown to improve outcomes by delivering synchronized electrical stimuli to the right and left ventricles utilizing an an endocardial right atrial lead, an endocardial right ventricular lead, and an epicardial left ventricular lead implanted in a branch of the coronary sinus.
  For LVEF≤35% a biventricular pacemaker-defibrillator will be implanted while for LVEF 36-50% a biventricular pacemaker will be implanted.
  Arms: Biventricular Pacing (BiVP)

SUMMARY:
The investigators aim to prospectively test the comparative effectiveness of His or Left bundle branch pacing in relation to patient centered outcomes (quality of life, physical activity, heart failure hospitalization, mortality) and comparative safety in relation to device-related complications and re-interventions (e.g., lead dislodgement, infection) relative to standard of care biventricular pacing in patients with heart failure due to left ventricular systolic dysfunction (LVEF≤50%) and with either a wide QRS (≥130 ms) or with/anticipated >40% pacing who are already receiving current standard heart failure pharmacological therapy.

DETAILED DESCRIPTION:
In this prospective, randomized, multi-center clinical trial, the investigators aim to prospectively evaluate the comparative effectiveness His or Left bundle branch pacing (His/LBBP) vs. biventricular pacing (BiVP) in patients with heart failure due to left ventricular systolic dysfunction (LVEF≤50%) and with either a wide QRS (≥130 ms) or with/anticipated >40% pacing who are already receiving current standard heart failure pharmacological therapy by assessing all cause death and heart failure hospitalization at the end of the study.

Additional formal secondary objectives include evaluation disease-specific quality and psychological adjustment changes at 1 year after device implant and evaluation of a composite of death of any cause or heart failure hospitalization or more >15% increase in the left ventricular end-systolic volume index at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age or older.
* A LVEF ≤ 50% within 6 months prior to enrollment.
* Resting QRS duration ≥130 ms as evidenced by a historical 12-lead ECG prior to enrollment OR anticipated right ventricular pacing >40% OR device in place with right ventricular pacing > 40%.
* Are optimized on HF guideline directed medical therapy according to current HF published guidelines OR patient's physician will make an effort to start all guideline-directed medical therapy and titrate doses up as permitted by the participant clinical status and co-morbidities prior to implantation procedure.

Exclusion Criteria:

* Women who are pregnant, lactating, or plan to become pregnant during the course of the trial.
* Participants with angiographic evidence of coronary disease who are candidates for coronary revascularization and are likely to undergo coronary artery bypass graft surgery or percutaneous coronary, intervention in the next three (3) months.
* Enzyme-positive myocardial infarction within the past three (3) months prior to enrollment.
* Coronary artery bypass graft surgery or percutaneous coronary intervention (balloon and/or stent angioplasty) within the past three (3) months prior to enrollment.
* Reversible non-ischemic cardiomyopathy (e.g., acute viral myocarditis).
* Participants with Chagas disease, cardiac sarcoidosis or amyloidosis.
* Expected to receive left ventricular assist device or heart transplantation within 6 months.
* Participants with primary severe valvular disease (e.g., aortic stenosis).
* Have a life expectancy of less than 12 months.
* Participants with irreversible brain damage from preexisting cerebral disease.
* Participants with a contrast dye allergy unable or unwilling to undergo pretreatment with steroids and/or diphenhydramine.
* Participants participating in any other interventional cardiovascular clinical trial.
* Participants who would be unable to comply with the study's follow-up visit schedule; or
* Participants who had any prior unsuccessful attempt at implantation of biventricular pacing (BiVP), His Bundle Pacing (HBP), or Left Bundle Branch Pacing (LBBP) device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2136 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
A combined clinical endpoint of all-cause mortality and hospitalization for heart failure | 5.5 years
  The primary efficacy outcome will be described using Kaplan-Meier freedom from event curves over time, with event-free survival compared between assigned treatment arms using a logrank test, stratified by levels of the two factors (LVEF (≤35% vs. 36 to 50%) and conduction abnormality (LBBB vs non-LBBB)) used for randomization.

SECONDARY OUTCOMES:
Assess change in Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) at 12 months | 12 months
  Assess change in Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) item score measured before and at 12 months after implant.
Change in composite endpoint comprised of death, first hospitalization for worsening HF and left ventricular end systolic volume index (LVESVi) at 5.5 years | 5.5 years
  Secondary endpoint measured from all cause death, first hospitalization for heart failure and echocardiography on left ventricular end-systolic volume index (LVESVi) in the His/LBBP vs. BIV-BiVP arm
Composite of cardiovascular death or heart transplant or durable left ventricular assist device or more > 15% increase in the LVESVi or change in KCCQ-12 at the end of the study using win ratio | 5.5 years
  Secondary endpoint measured from cardiovascular death or heart transplant or durable left ventricular assist device or more > 15% increase in the LVESVi or change in KCCQ-12 at the end of the study using win ratio
Death from any cause at 5.5 years | 5.5 years
  Secondary endpoint measured from all cause death
Death from any cardiovascular cause at 5.5 years | 5.5 years
  Secondary endpoint measured from death due to cardiovascular causes
Hospitalization for heart failure at 5.5 years | 5.5 years
  Secondary endpoint measured from first hospitalization for heart failure
Cardiovascular hospitalization at 5.5 years | 5.5 years
  Secondary endpoint measured from first hospitalization for cardiovascular disease
Total HF hospitalizations | 5.5 years
  Total number of HF hospitalizations
Composite of cardiovascular death or first HF hospitalization | 5.5 years
  Secondary endpoint measured from cardiovascular death, first hospitalization for heart failure
Composite cardiovascular death or HF hospitalization or heart transplant or durable left ventricular assist device | 5.5 years
  Secondary endpoint measured from cardiovascular death, heart transplant or durable left ventricular assist device
Change in NYHA Classification at 12 months | 12 months
  Secondary endpoint measured from New York Heart Association class
Change in Six Minute Walk Test performance at 12 months | 12 months
  Secondary endpoint measured from Six Minute Walk Test
Patient activity measured through cardiovascular implantable electronic devices (CIED) at 12 months | 12 months
  Measurement Patient activity measured through cardiovascular implantable electronic devices (CIED)
Change in NT-proBNP at 12 months | 12 months
  Measurement of heart failure serum biomarker NT-proBNP

OTHER OUTCOMES:
Appropriate ICD therapy for ventricular arrhythmias | 5.5 years
  Antitachycardia pacing or ICD shocks
Incidence of atrial tachyarrhythmia events | 5.5 years
  Atrial arrhythmia event measured through cIED
Change in Left Ventricular Ejection Fraction (LVEF) at 12 months | 12 months
  Measurement of LVEF before and at 12 months after implant using echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Mihail G Chelu, MD, PhD, Principal Investigator — Baylor College of Medicine; Kenneth A Ellenbogen, MD, Principal Investigator — Virginia Commonwealth University
Locations (71):
- United States (57):
  - Mercy Gilbert & Chandler Regional Medical Centers, Gilbert AZ, Gilbert, Arizona
  - University of Arizona College of Medicine- Phoenix, Tucson, Arizona
  - University of Arkansas for Medical Sciences (UAMS), Little Rock, Arkansas
  - University of California San Diego, La Jolla, California
  - University of Colorado (Anschutz Medical Campus), Denver, Colorado
  - South Denver Cardiology Associates, Littleton, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Heart Rhythm Solutions, Davie, Florida
  - University of Florida Jacksonville, Jacksonville, Florida
  - Mount Sinai Medical Center of Florida, Inc., Miami Beach, Florida
  - Cleveland Clinic Florida, Palm Beach Gardens, Florida
  - Florida Heart and Vascular, LLC dba Florida Heart Rhythm Specialist, PLLC, South Pasadena, Florida
  - University of South Florida, Tampa, Florida
  - Rush University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - CIS Clinical Research Corporation, Naperville, Illinois
  - Trustees of Indiana University, Indianapolis, Indiana
  - Baptist Health Louisville, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - HMH Hospitals Corporation, Hackensack, New Jersey
  - Virtua Health, Marlton, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - The Valley Hospital, Inc., Ridgewood, New Jersey
  - Lovelace Medical Center, Albuquerque, New Mexico
  - Weill Cornell Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center/New York-Presbyterian Hospital (CUMC/NYPH), New York, New York
  - MH Mission Hospital LLLP- Asheville Cardiology Associates, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Novant Health, Charlotte, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - The MetroHealth System, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - St. Luke's University Health Network, Allentown, Pennsylvania
  - Lehigh Valley Hospital Inc., Allentown, Pennsylvania
  - Penn Medicine Lancaster General, Lancaster, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - University of Pittsburg, Pittsburgh, Pennsylvania
  - Geisinger Commonwealth School of Medicine, Scranton, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Prisma Health-Upstate, Greenville, South Carolina
  - Texas Health Research & Education Institute, Arlington, Texas
  - Baylor College of Medicine, Houston, Texas
  - St. Mark's Hospital, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - Inova Heart and Vascular Institute, Falls Church, Virginia
  - Sentara Healthcare, Newport News, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
- Canada (14):
  - Mazankowski Alberta Heart Institute/University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Victoria Cardiac Arrhythmia Trials (VCAT) Inc., Victoria, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Hamilton Health Sciences (HHS), Hamilton, Ontario
  - Newmarket Electrophysiology Research Group Inc. (NERG), Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - CIUSSS de l'Estrie - CHUS, Saint-Jean-sur-Richelieu, Quebec
  - University of Calgary, Calgary
  - Waterloo Wellington Cardiovascular Research Institute (WWCRI) - St. Mary's General Hospital, Kitchener
  - Research Institute of the McGill University Health Centre (RI-MUHC) - MUHC, Montreal General Hospital, Montreal
  - Université Laval, Québec

IPD SHARING:
Plan to Share IPD: No